CLINICAL TRIAL: NCT00295542
Title: Prognostic Value of Ambulatory Blood Pressure Monitoring in the Prediction of Cardiovascular Events and Effects of Chronotherapy in Relation to Risk (the MAPEC Study).
Brief Title: Ambulatory Blood Pressure Monitoring in the Prediction of Cardiovascular Events and Effects of Chronotherapy
Acronym: MAPEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other); Ministry of Work and Welfare - Xunta de Galicia (Other Government); Ministerio de Educacion y Ciencia, Spain (Unknown)
Responsible Party: Ramon C. Hermida, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGIDIT03-PXIB-32201PR; SAF2006-6254; INCITE07-PXI-322003ES
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Hypertension
Keywords: ambulatory blood pressure monitoring; cardiovascular risk; chronotherapy; circadian pattern
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure Monitoring, Ambulatory; Chronotherapy; Angiotensin-Converting Enzyme Inhibitors; Enalapril; Quinapril; Lisinopril; Telmisartan; olmesartan; Adrenergic beta-Antagonists; Atenolol; Carvedilol; Diuretics; Torsemide; Indapamide; Doxazosin; Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment on awakening
  Interventions: Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of antihypertensive medication; Drug: ACEI (including spirapril, enalapril, quinapril, lisinopril); Drug: ARB (including valsartan, telmisartan, olmesartan); Drug: beta blockers (including nebivolol, atenolol, carvedilol); Drug: diuretics (torasemide, indapamide, HTCZ) and doxazosin; Procedure: Combination therapy in essential hypertension
- 2 (Active Comparator): Treatment at bedtime
  Interventions: Device: Ambulatory blood pressure monitoring; Procedure: Chronotherapy, timing of antihypertensive medication; Drug: ACEI (including spirapril, enalapril, quinapril, lisinopril); Drug: ARB (including valsartan, telmisartan, olmesartan); Drug: beta blockers (including nebivolol, atenolol, carvedilol); Drug: diuretics (torasemide, indapamide, HTCZ) and doxazosin; Procedure: Combination therapy in essential hypertension

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring — Sampling at 20-min intervals from 07:00 to 23:00 hours and at 30-min intervals at night for 48 consecutive hours
Procedure: Chronotherapy, timing of antihypertensive medication — Comparison of effects of awakening versus bedtime dosing
Drug: ACEI (including spirapril, enalapril, quinapril, lisinopril) — Treatment at awakening versus bedtime
Drug: ARB (including valsartan, telmisartan, olmesartan) — Treatment at awakening versus bedtime
Drug: beta blockers (including nebivolol, atenolol, carvedilol) — Treatment at awakening versus bedtime
Drug: diuretics (torasemide, indapamide, HTCZ) and doxazosin — Treatment at awakening versus bedtime
Procedure: Combination therapy in essential hypertension — Treatment at awakening versus bedtime

SUMMARY:
The MAPEC study was designed to investigate whether normalizing the circadian blood pressure profile towards a more dipper pattern (increasing the diurnal/nocturnal ratio of blood pressure) by the use of Chronotherapy (that is, taking into account the time of day of administration of antihypertensive medications) reduces cardiovascular risk.

DETAILED DESCRIPTION:
Target organ damage is more closely associated with ambulatory (ABPM) than with clinic blood pressure (BP). In particular, the reduction of the normal 10 to 20% sleep-time BP decline (non-dipper pattern) is associated with elevated risk of end-organ injury, particularly to the heart, brain and kidney. These results suggest that cardiovascular risk could be influenced not by BP elevation alone, but also by the magnitude of the circadian BP variability. Moreover, at least two independent prospective studies have suggested that nighttime BP is a better predictor of risk than daytime BP. Common to all previous trials is that prognostic significance of ABPM has relied on a single baseline profile from each participant, without accounting for possible changes in the BP pattern, mainly associated to antihypertensive therapy and aging during follow-up. The MAPEC study investigates, first, the comparative prognostic value of several BP parameters (including, among many others, BP variability, the diurnal/nocturnal ratio, diurnal and nocturnal means, slope of morning rise, etc) in the prediction of cardiovascular morbidity and mortality; and, second, whether potential changes in the circadian BP pattern after Chronotherapy with antihypertensive drugs are associated to changes in cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension

Exclusion Criteria:

* AIDS
* shift workers
* secondary hypertension
* intolerant to ABPM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3344 (Actual)
Dates: Start 2000-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Prognostic value of ABPM, impact of changes in ambulatory BP and impact of circadian time of antihypertensive treatment in cardiovascular, cerebrovascular and renal risk assessment. | Five years

SECONDARY OUTCOMES:
Influence of circadian time of antihypertensive treatment in BP control and the remodeling of the circadian BP pattern of hypertensive patients. | Five years
Prevalence of an altered BP profile as a function of the circadian time of treatment. | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Ramon C Hermida, PhD, Principal Investigator — University of Vigo
Locations (1):
- Hospital Clinico Universitario, Santiago de Compostela, Spain

REFERENCES:
- [Derived] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Bedtime ingestion of hypertension medications reduces the risk of new-onset type 2 diabetes: a randomised controlled trial. Diabetologia. 2016 Feb;59(2):255-65. doi: 10.1007/s00125-015-3749-7. Epub 2015 Sep 23. PMID 26399404
- [Derived] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Decreasing sleep-time blood pressure determined by ambulatory monitoring reduces cardiovascular risk. J Am Coll Cardiol. 2011 Sep 6;58(11):1165-73. doi: 10.1016/j.jacc.2011.04.043. PMID 21884956
- [Derived] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Influence of time of day of blood pressure-lowering treatment on cardiovascular risk in hypertensive patients with type 2 diabetes. Diabetes Care. 2011 Jun;34(6):1270-6. doi: 10.2337/dc11-0297. PMID 21617110
- [Derived] Hermida RC, Ayala DE, Mojon A, Fernandez JR. Ambulatory blood pressure control with bedtime aspirin administration in subjects with prehypertension. Am J Hypertens. 2009 Aug;22(8):896-903. doi: 10.1038/ajh.2009.83. Epub 2009 Apr 30. PMID 19407805